CLINICAL TRIAL: NCT01251796
Title: A Phase I Study of ARQ 197 in Combination With Erlotinib in CYP2C19 Poor Metabolizer Patients With Advanced/Recurrent Non-Small-Cell Lung Cancer
Brief Title: A Study of ARQ 197 in Combination With Erlotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: ARQ 197-005
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Advanced/Recurrent Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197; Erlotinib Hydrochloride

ARMS (1):
- ARQ 197 and Erlotinib (Experimental): ARQ 197 and erlotinib hydrochloride
  Interventions: Drug: ARQ 197 and Erlotinib

INTERVENTIONS:
Drug: ARQ 197 and Erlotinib — Orally twice daily administration of ARQ197 and orally once daily administration of erlotinib hydrochloride

SUMMARY:
This is a phase I study to determine the safety, tolerability and recommended phase II dose of ARQ 197 given in combination with erlotinib as primary endpoints in CYP2C19 poor metabolizer patients with advanced/recurrent non-small-cell lung cancer. The pharmacokinetic profile and antitumor activity of ARQ 197 administered alone or in combination with erlotinib will also be determined as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent for study participation must be obtained
* A histologically or cytologically confirmed advanced/recurrent non-small-cell lung cancer
* History of ≥1 prior chemotherapy regimen (treatment with EGFR tyrosine kinase inhibitors will be counted as one regimen)
* ECOG PS of 0 or 1
* Life expectancy of ≥3 months
* Poor metabolizers as defined by CYP2C19 genotype

Exclusion Criteria:

* Anti-cancer chemotherapy, anti-cancer therapy with EGFR-TKI, hormone therapy, radiotherapy, immunotherapy, other investigational agents or anti-cancer antibody therapy within 28 days prior to ARQ 197 dose
* Surgery for cancer within 28 days prior to ARQ 197 dose
* Active double cancer
* Known symptomatic brain metastases
* An intercurrent illness that is uncontrolled (e.g., infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic arrhythmia, interstitial pneumonia)
* Pregnant or lactating
* Subjects who wish to have a child and who would not agree to use contraceptive measures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity in the combination of tivantinib and erlotinib | DLT observation period started from the day of first single agent treatment to the day after the continuous combination treatment for 29 days.
  Tivantinib was treated once as a single agent on Day 1. After 2 days of interruption, dayly treatments of the combination started.

SECONDARY OUTCOMES:
Pharmacokinetic profile of ARQ 197 | Plasma sample correction at pre-dose, 1, 2, 4, 6, 10, 12 and 24 hours on Day 1, and in addition, at pre-dose, 1, 2, 4, 6, 10, 12 hours on the day of the first comnibation treatment
  Summary statistics of plasma concentration and pharmacokinetic parameters
Pharmacokinetic profile of Erlotinib | At pre-dose, 1, 2, 4, 6, 10, 12 hours on the day of the first comnibation treatment
  Summary statistics of plasma concentration and pharmacokinetic parameters
Antitumor activity | Baseline, and then every 6 week of imaging until discontinuation criteria met
  Response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shizuoka, Japan